CLINICAL TRIAL: NCT04195750
Title: An Open-label, Randomized Phase 3 Study of MK-6482 Versus Everolimus in Participants With Advanced Renal Cell Carcinoma That Has Progressed After Prior PD-1/L1 and VEGF-Targeted Therapies
Brief Title: A Study of Belzutifan (MK-6482) Versus Everolimus in Participants With Advanced Renal Cell Carcinoma (MK-6482-005)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482-005; MK-6482 (Other: MSD); 205262 (Registry Identifier: Japic-CTI); jRCT2080225166 (Other: jRCT); 2023-506635-15 (Registry Identifier: EU CT); U1111-1294-1321 (Registry Identifier: UTN); 2019-003444-72 (EudraCT Number)
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma, Renal Cell
Keywords: Hypoxia inducible Factor (HIF); Hypoxia inducible factor 1B (HIF-1B); Hypoxia inducible factor 2 alpha (HIF-2 alpha); Hypoxia inducible factor 2α (HIF-2α); Renal Cell Carcinoma (RCC); Kidney Cancer; PT-2977; PT2977; MK6482
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — belzutifan; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Belzutifan (Experimental): Randomized participants received 120 mg of belzutifan orally once daily (QD), until disease progression or discontinuation.
  Interventions: Drug: Belzutifan
- Everolimus (Active Comparator): Randomized participants received 10 mg of Everolimus orally QD, until disease progression or discontinuation.
  Interventions: Drug: Everolimus
- Safety Run-In (Experimental): Non-Randomized participants enrolled into the Safety Run-in received up to 120 mg of belzutifan QD.
  Interventions: Drug: Belzutifan

INTERVENTIONS:
Drug: Belzutifan — Oral tablets
  Other Names: MK-6482; WELIREG™
  Arms: Belzutifan; Safety Run-In
Drug: Everolimus — Oral tablets
  Other Names: Afinitor; Afinitor DISPERZ; Zortress
  Arms: Everolimus

SUMMARY:
The primary objective of this study is to compare belzutifan to everolimus with respect to progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR) and to compare everolimus with respect to overall survival (OS). The hypothesis is that belzutifan is superior to everolimus with respect to PFS and OS.

DETAILED DESCRIPTION:
Per protocol, all participants enrolled in the Safety Run-In were not randomized and not included in the protocol-specified analyses for any of the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Has unresectable, locally advanced or metastatic clear cell renal cell carcinoma (RCC)
* Has had disease progression on or after having received systemic treatment for locally advanced or metastatic RCC with both Programmed cell death 1 ligand 1 (PD-1/L1) checkpoint inhibitor and a vascular endothelial growth factor - tyrosine kinase inhibitor (VEGF-TKI) in sequence or in combination
* Has received no more than 3 prior systemic regimens for locally advanced or metastatic RCC
* A male participant is eligible to participate if he is abstinent from heterosexual intercourse or agrees to use contraception during the intervention period and for at least 7 days after the last dose of study intervention
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies: Not a woman of childbearing potential (WOCBP) OR a WOCBP who agrees to follow the contraceptive guidance during the intervention period and for at least 30 days after the last dose of study intervention for those randomized to belzutifan and for at least 8 weeks after the last dose of study intervention for those randomized to everolimus
* The participant (or legally acceptable representative if applicable) has provided documented informed consent for the study
* Has adequate organ function

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. (Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ [e.g., breast carcinoma, cervical cancer in situ] that have undergone potentially curative therapy are not excluded)
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis. (Participants with previously treated brain metastases may participate provided they are radiologically stable for at least 4 weeks (28 days) by repeat imaging)
* Has clinically significant cardiac disease, including unstable angina, acute myocardial infarction within 6 months from Day 1 of study medication administration, or New York Heart Association Class III or IV congestive heart failure. (Medically controlled arrhythmia stable on medication is permitted)
* Has poorly controlled hypertension defined as systolic blood pressure (SBP) ≥150 mm Hg and/or diastolic blood pressure (DBP) ≥90 mm Hg
* Has moderate to severe hepatic impairment (Child-Pugh B or C)
* Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study
* Is unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption (e.g., gastrectomy, partial bowel obstruction, malabsorption)
* Has known hypersensitivity or allergy to the active pharmaceutical ingredient or any component of the study intervention (belzutifan or everolimus) formulations
* Has received prior treatment with belzutifan or another hypoxia inducible factor 2α (HIF-2α inhibitor)
* Has received prior treatment with everolimus or any other specific or selective target of rapamycin complex 1 (TORC1)/ phosphatidylinositol 3-kinase (PI3K)/ protein kinase B (AKT) inhibitor (e.g., temsirolimus) in the advanced disease setting
* Has received any type of systemic anticancer antibody (including investigational antibody) within 4 weeks before randomization
* Has received prior radiotherapy within 2 weeks prior to randomization
* Has had major surgery within 3 weeks prior to randomization
* Has received a live vaccine within 30 days prior to randomization. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines are live attenuated vaccines and are not allowed
* Is currently receiving either strong (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil) inhibitors of cytochrome P450 3A4 (CYP3A4) that cannot be discontinued for the duration of the study
* Is currently receiving either strong (phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate (e.g., bosentan, efavirenz, modafinil) inducers of CYP3A4 that cannot be discontinued for the duration of the study
* Is currently participating in a study of an investigational agent or is currently using an investigational device
* Has an active infection requiring systemic therapy
* Has active bacillus tuberculosis (TB)
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to randomization
* Has a known history of human immunodeficiency virus (HIV) infection. (Testing for HIV at screening is only required if mandated by local health authority
* Has a known history of Hepatitis B virus (HBV) (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (HCV) (defined as HCV ribonucleic acid [RNA] [qualitative] is detected) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2026-09-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (172):
- United States (29):
  - University of Alabama - Birmingham ( Site 1538), Birmingham, Alabama
  - University of California San Diego Moores Cancer Center ( Site 1546), La Jolla, California
  - St Joseph Heritage Healthcare ( Site 1531), Santa Rosa, California
  - University Of Colorado ( Site 1540), Aurora, Colorado
  - UCHealth Highlands Ranch Hospital ( Site 1560), Highlands Ranch, Colorado
  - Sibley Memorial Hospital ( Site 1559), Washington D.C., District of Columbia
  - Northwest Georgia Oncology Centers PC ( Site 1520), Marietta, Georgia
  - The University of Chicago Medical Center ( Site 1539), Chicago, Illinois
  - Ochsner Medical Center ( Site 1522), New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins ( Site 1514), Baltimore, Maryland
  - Massachusetts General Hospital ( Site 1558), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center ( Site 1501), Boston, Massachusetts
  - Dana Farber Cancer Institute ( Site 1505), Boston, Massachusetts
  - Henry Ford Cancer Center ( Site 1511), Detroit, Michigan
  - Hattiesburg Clinic ( Site 1509), Hattiesburg, Mississippi
  - St. Vincent Frontier Cancer Center ( Site 1549), Billings, Montana
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 1513), Hackensack, New Jersey
  - University of Rochester Medical Center ( Site 1543), Rochester, New York
  - University of North Carolina at Chapel Hill ( Site 1537), Chapel Hill, North Carolina
  - Oncology Hematology Care, Inc. ( Site 1524), Cincinnati, Ohio
  - Cleveland Clinic ( Site 1504), Cleveland, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC ( Site 1523), Tulsa, Oklahoma
  - Oregon Health & Science University ( Site 1553), Portland, Oregon
  - Abramson Cancer Center ( Site 1525), Philadelphia, Pennsylvania
  - Fox Chase Cancer Center ( Site 1506), Philadelphia, Pennsylvania
  - Medical University of South Carolina ( Site 1518), Charleston, South Carolina
  - Henry Joyce Cancer Clinic ( Site 1544), Nashville, Tennessee
  - Texas Oncology-Austin Central ( Site 1533), Austin, Texas
  - Texas Oncology, P.A.-Dallas ( Site 1534), Dallas, Texas
- Brazil (5):
  - Centro Avancado de Tratamento Oncologico ( Site 1657), Belo Horizonte, Minas Gerais
  - Instituto de Cancer e Transplante de Curitiba ICTR ( Site 1650), Curitiba, Paraná
  - Liga Norte Riograndense Contra o Cancer ( Site 1651), Natal, Rio Grande do Norte
  - Hospital de Clinicas de Porto Alegre ( Site 1655), Porto Alegre, Rio Grande do Sul
  - Real e Benemerita Associacao Portuguesa de Beneficencia ( Site 1653), São Paulo
- Canada (6):
  - BC Cancer - Vancouver Center ( Site 0155), Vancouver, British Columbia
  - Nova Scotia Health Authority QEII-HSC ( Site 0150), Halifax, Nova Scotia
  - Juravinski Cancer Centre ( Site 0154), Hamilton, Ontario
  - Sunnybrook Research Institute ( Site 0153), Toronto, Ontario
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0151), Montreal, Quebec
  - CHUQ-Univ Laval-Hotel Dieu de Quebec ( Site 0152), Québec, Quebec
- Chile (2):
  - Bradfordhill ( Site 0003), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 0004), Temuco, Región de la Araucanía
- Colombia (5):
  - Fundacion Centro de Investigacion Clinica CIC ( Site 1703), Medellín, Antioquia
  - Administradora Country SA - Clinica del Country ( Site 1701), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 1709), Valledupar, Cesar Department
  - Clinica Colsanitas S.A. Sede Clinica Universitaria Colombia ( Site 1702), Bogota, Cundinamarca
  - Oncologos del Occidente S.A. ( Site 1708), Pereira, Risaralda Department
- Czechia (6):
  - Masarykuv onkologicky ustav ( Site 0105), Brno, Brno-mesto
  - Fakultni nemocnice Ostrava ( Site 0103), Ostrava, Ostrava Mesto
  - Fakultni nemocnice Hradec Kralove ( Site 0106), Hradec Králové
  - Fakultni nemocnice Olomouc ( Site 0104), Olomouc
  - Fakultni nemocnice Kralovske Vinohrady ( Site 0102), Prague
  - Fakultni Thomayerova nemocnice ( Site 0107), Prague
- Denmark (2):
  - Herlev Hospital ( Site 0251), Herlev, Capital Region
  - Aarhus University Hospital Skejby ( Site 0250), Aarhus, Central Jutland
- Finland (4):
  - Kuopion Yliopistollinen Sairaala ( Site 0304), Kuopio, Northern Savonia
  - Tampereen yliopistollinen sairaala ( Site 0300), Tampere, Pirkanmaa
  - TYKS T-sairaala Syopatautien pkl ( Site 0301), Turku, Southwest Finland
  - HYKS. ( Site 0302), Helsinki, Uusimaa
- France (8):
  - CHU de Bordeaux Hop St ANDRE ( Site 0359), Bordeaux, Aquitaine
  - Institut de cancérologie Strasbourg Europe (ICANS) ( Site 0350), Strasbourg, Bas-Rhin
  - Centre Francois Baclesse ( Site 0360), Caen, Calvados
  - CHU Besancon - Hopital Jean Minjoz ( Site 0351), Besançon, Doubs
  - Institut de Cancerologie du Gard - CHU Caremeau ( Site 0352), Nîmes, Gard
  - Centre Alexis Vautrin Institut de Cancerologie de Lorraine ( Site 0356), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Centre Hospitalier Lyon Sud ( Site 0354), Pierre-Bénite, Rhone
  - Gustave Roussy ( Site 0353), Villejuif, Val-de-Marne
- Germany (8):
  - Universitaetsklinik fuer Urologie ( Site 0405), Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Duesseldorf ( Site 0410), Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Essen ( Site 0401), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden ( Site 0403), Dresden, Saxony
  - Universitaetsklinikum Magdeburg A.o.R. ( Site 0404), Magdeburg, Saxony-Anhalt
  - Universitaetsklinikum Jena ( Site 0402), Jena, Thuringia
  - Universitaetsmedizin Berlin ( Site 0400), Berlin
  - Universitatsklinikum Hamburg-Eppendorf ( Site 0408), Hamburg
- Hong Kong (4):
  - Prince of Wales Hospital ( Site 1050), Hong Kong
  - Queen Mary Hospital ( Site 1051), Hong Kong
  - Queen Elizabeth Hospital. ( Site 1052), Kowloon
  - Princess Margaret Hospital. ( Site 1053), Lai Chi Kok
- Hungary (6):
  - Bekes Megyei Kozponti Korhaz - Pandy Kalman Tagkorhaza ( Site 0505), Gyula, Bekes County
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Okta-Klinikai Onkológiai és Sugárterápiás Ce, Miskolc, Borsod-Abauj Zemplen county
  - Semmelweis Egyetem ( Site 0501), Budapest
  - Orszagos Onkologiai Intezet ( Site 0503), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 0504), Debrecen
  - Zala Megyei Szent Rafael Korhaz ( Site 0509), Zalaegerszeg
- Italy (10):
  - Istituto Oncologico Veneto IRCCS ( Site 0603), Padua, Veneto
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento-Oncology Unit ( Site 0605, Verona, Veneto
  - Medical Oncology Ospedale San Donato ( Site 0609), Arezzo
  - Azienda Ospedaliera Policlinico di Bari ( Site 0610), Bari
  - Policlinico S. Orsola-Malpighi ( Site 0606), Bologna
  - Istituto Nazionale dei Tumori ( Site 0601), Milan
  - Azienda Ospedaliero Universitaria di Modena Policlinico ( Site 0604), Modena
  - Fondazione Salvatore Maugeri clinica del lavoro ( Site 0600), Pavia
  - Fondazione Policlinico Universitario A. Gemelli ( Site 0607), Roma
  - Azienda Ospedaliera Santa Maria ( Site 0602), Terni
- Japan (23):
  - Fujita Health University ( Site 1016), Toyoake, Aichi-ken
  - National Cancer Center Hospital East ( Site 1001), Kashiwa, Chiba
  - Ehime University Hospital ( Site 1014), Tōon, Ehime
  - Sapporo Medical University Hospital ( Site 1008), Sapporo, Hokkaido
  - Yokohama City University Hospital ( Site 1015), Yokohama, Kanagawa
  - Kanagawa cancer center ( Site 1021), Yokohama, Kanagawa
  - Nara Medical University Hospital ( Site 1009), Kashihara, Nara
  - Kindai University Hospital- Osakasayama Campus-Urology ( Site 1011), Sayama, Osaka
  - Osaka University Hospital ( Site 1006), Suita, Osaka
  - Saitama Medical University International Medical Center ( Site 1012), Hidaka, Saitama
  - Hamamatsu University Hospital ( Site 1005), Hamamatsu, Shizuoka
  - Toyama University Hospital ( Site 1013), Toyoma, Toyama
  - Yamaguchi University Hospital ( Site 1018), Ube, Yamaguchi
  - Kyushu University Hospital ( Site 1007), Fukuoka
  - Hiroshima University Hospital-Hiroshima University Hospital ( Site 1019), Hiroshima
  - Niigata University Medical & Dental Hospital ( Site 1022), Niigata
  - Okayama University Hospital ( Site 1020), Okayama
  - Tokushima University Hospital-Department of Urology ( Site 1017), Tokushima
  - National Cancer Center Hospital ( Site 1003), Tokyo
  - Toranomon Hospital ( Site 1004), Tokyo
  - Nippon Medical School Hospital ( Site 1010), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 1000), Tokyo
  - Keio University Hospital ( Site 1002), Tokyo
- Norway (2):
  - Akershus universitetssykehus ( Site 0851), Lorenskog, Akershus
  - Helse Bergen HF - Haukeland Universitetssykehus ( Site 0854), Bergen, Hordaland
- Russia (11):
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 1151), Krasnoyarsk, Krasnoyarsk Krai
  - SBIH City clinical hospital named after D.D. Pletniov ( Site 1160), Moscow, Moscow
  - N.N. Blokhin NMRCO ( Site 1156), Moscow, Moscow
  - Russian Scientific Center of Roentgenoradiology ( Site 1155), Moscow, Moscow
  - First Moscow State Medical University n.a. I.M.Sechenov ( Site 1163), Moscow, Moscow
  - Central Clinical Hospital with Polyclinic ( Site 1157), Moscow, Moscow
  - Hadassah Medical-Oncology department ( Site 1164), Moscow, Moscow Oblast
  - Omsk Clinical Oncology Dispensary ( Site 1150), Omsk, Omsk Oblast
  - Russian Scientific Center of Radiology and Surgical Technologies ( Site 1153), Saint Petersburg, Sankt-Peterburg
  - SBHI SPb Clinical Research Centre of specialized types of medical care ( Site 1159), Saint Petersburg, Sankt-Peterburg
  - City clinical oncological dispensary ( Site 1154), Saint Petersburg, Sankt-Peterburg
- South Korea (6):
  - National Cancer Center ( Site 1204), Gyeonggi-do, Kyonggi-do
  - Chungnam National University Hospital ( Site 1205), Daejeon, Taejon-Kwangyokshi
  - Korea University Anam Hospital ( Site 1203), Seoul
  - Severance Hospital Yonsei University Health System ( Site 1202), Seoul
  - Asan Medical Center ( Site 1200), Seoul
  - Samsung Medical Center ( Site 1201), Seoul
- Spain (5):
  - Instituto Catalan de Oncologia - ICO ( Site 1251), L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Vall d Hebron ( Site 1250), Barcelona, Catalonia
  - Hospital General Universitario 12 de Octubre ( Site 1252), Madrid, Madrid, Comunidad de
  - Instituto Valenciano de Oncologia - IVO ( Site 1254), Valencia, Valenciana, Comunitat
  - Hospital Ramon y Cajal ( Site 1253), Madrid
- Sweden (4):
  - Laenssjukhuset Ryhov ( Site 1853), Jönköping, Jönköping County
  - Malmo Universitetssjukhus ( Site 1851), Malmo, Skåne County
  - Karolinska Universitetssjukhuset Solna ( Site 1850), Stockholm, Stockholm County
  - Norrlands Universitetssjukhus ( Site 1856), Umeå, Västerbotten County
- Taiwan (6):
  - Chang Gung Medical Foundation - Kaohsiung ( Site 1104), Kaohsiung City
  - Taichung Veterans General Hospital ( Site 1105), Taichung
  - National Cheng Kung University Hospital ( Site 1103), Tainan
  - National Taiwan University Hospital ( Site 1100), Taipei
  - Taipei Veterans General Hospital ( Site 1101), Taipei
  - Chang Gung Medical Foundation-Linkou Branch-Urology ( Site 1106), Taoyuan District
- Turkey (Türkiye) (8):
  - Ankara Universitesi Tip Fakultesi ( Site 1311), Ankara
  - Hacettepe Universitesi Tip Fakultesi ( Site 1300), Ankara
  - Gazi Universitesi Tip Fakultesi ( Site 1308), Ankara
  - Trakya University Medical Faculty Balkan Oncology Hospital ( Site 1302), Edirne
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 1305), Istanbul
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 1303), Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi ( Site 1304), Izmir
  - Izmir Katip Celebi Universitesi Ataturk Egitim ve Arastirma Hastanesi ( Site 1306), Izmir
- Ukraine (3):
  - MI Dnipr Regional Clinical Hospital named after I.I. Mechnikov ( Site 1453), Dnipropetrovsk, Dnipropetrovsk Oblast
  - MI Precarpathian Clinical Oncology Center ( Site 1452), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Kyiv City Clinical Oncology Center ( Site 1450), Kyiv, Kyivska Oblast
- United Kingdom (9):
  - Cambridge University Hospitals NHSFT ( Site 1405), Cambridge, Cambridgeshire
  - Western General Hospital ( Site 1400), Edinburgh, Edinburgh, City of
  - The Beatson West of Scotland Cancer Centre ( Site 1402), Glasgow, Glasgow City
  - Barts Health NHS Trust ( Site 1407), London, London, City of
  - Royal Marsden NHS Foundation Trust ( Site 1403), London, London, City of
  - Imperial Healthcare NHS Trust Charing Cross Hospital ( Site 1409), London, London, City of
  - Royal Marsden Hospital Sutton-Surrey ( Site 1411), Sutton, Surrey
  - Medway Maritime Hospital ( Site 1406), Gillingham
  - The Christie NHS Foundation Trust ( Site 1401), Manchester

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Choueiri TK, Powles T, Peltola K, de Velasco G, Burotto M, Suarez C, Ghatalia P, Iacovelli R, Lam ET, Verzoni E, Gumus M, Stadler WM, Kollmannsberger C, Melichar B, Venugopal B, Gross-Goupil M, Poprach A, De Santis M, Schutz FA, Park SH, Nosov DA, Porta C, Lee JL, Garcia-Del-Muro X, Biscaldi E, Manneh Kopp R, Oya M, He L, Wang A, Perini RF, Vickery D, Albiges L, Rini B; LITESPARK-005 Investigators. Belzutifan versus Everolimus for Advanced Renal-Cell Carcinoma. N Engl J Med. 2024 Aug 22;391(8):710-721. doi: 10.1056/NEJMoa2313906. PMID 39167807
- [Derived] Powles T, Choueiri TK, Albiges L, Peltola K, de Velasco G, Burotto M, Suarez C, Ghatalia P, Iacovelli R, Lam ET, Verzoni E, Gumus M, Stadler WM, Kollmannsberger C, Melichar B, Venugopal B, Gross-Goupil M, Poprach A, De Santis M, Rizzo M, Shinde R, Saretsky TL, He L, Perini RF, Vickery D, Rini B. Health-related quality of life with belzutifan versus everolimus for advanced renal cell carcinoma (LITESPARK-005): patient-reported outcomes from a randomised, open-label, phase 3 trial. Lancet Oncol. 2025 Apr;26(4):491-502. doi: 10.1016/S1470-2045(25)00032-4. Epub 2025 Mar 17. PMID 40112850
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26230&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per protocol, the 9 participants enrolled in the Safety Run-In were not randomized and not included in the protocol-specified analyses for any of the outcome measures.
Period: Overall Study
Arm/Group | Belzutifan | Everolimus | Safety Run-In
Started | 374 | 372 | 9
Treated | 372 | 360 | 9
Completed | 0 | 0 | 0
Not Completed | 374 | 372 | 9
Not completed — Death | 245 | 253 | 5
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 9 | 8 | 0
Not completed — Ongoing | 120 | 110 | 4

BASELINE CHARACTERISTICS:
Population: Per protocol, the 9 participants enrolled in the Safety Run-In were not randomized and not included in the protocol-specified analyses for any of the outcome measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Belzutifan | Everolimus | Safety Run-In | Total
Number analyzed (Participants) | 374 | 372 | 9 | 755
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (10.2) | 63.1 (9.7) | 70.0 (6.6) | 62.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 88 | 4 | 169
  Male | 297 | 284 | 5 | 586
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 37 | 0 | 78
  Not Hispanic or Latino | 300 | 303 | 9 | 612
  Unknown or Not Reported | 33 | 32 | 0 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 0 | 5
  Asian | 43 | 47 | 9 | 99
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 4 | 4 | 0 | 8
  White | 297 | 291 | 0 | 588
  More than one race | 6 | 11 | 0 | 17
  Unknown or Not Reported | 21 | 16 | 0 | 37
International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) Risk Category [Count of Participants; unit: Participants] — Stratification factor per case report form based on the following risk factors: baseline Karnofsky Performance Status <80%; interval between initial diagnosis of renal cell carcinoma to start of first-line systemic treatment for advanced disease <1year; baseline hemoglobin <lower limit of normal (LLN); baseline platelet count >upper limit of normal (ULN); baseline corrected serum calcium >ULN; and baseline neutrophil >ULN. The category was determined by totaling the risk factors per participant: favorable (0 factors); intermediate (1-2 factors); and poor (≥3 factors).
  Participants
    Favorable | 81 | 84 | 6 | 171
    Intermediate | 248 | 242 | 3 | 493
    Poor | 45 | 46 | 0 | 91
Number of Prior Vascular Endothelial Growth Factor (VEGF)/VEGF-Receptor Targeted Therapies [Count of Participants; unit: Participants] — Stratification factor per case report form, the number of prior VEGF/VEGF-Receptor targeted therapies that they received to treat their advanced Renal Cell Carcinoma (RCC): 1 versus 2-3.
  Participants
    1 | 186 | 190 | 3 | 379
    2-3 | 188 | 182 | 6 | 376

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review is presented here.
Time Frame: Up to approximately 39 months
Population: Per protocol, the analysis population consisted of all randomized participants based on the treatment group to which they were randomized. Per protocol, participants enrolled in the Safety Run-In were not randomized and not included in the protocol-specified analyses for any of the outcome measures.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belzutifan | Everolimus
Number analyzed (Participants) | 374 | 372
Months | 5.6 [3.8 to 6.5] | 5.6 [4.8 to 5.8]
Statistical Analysis 1: Comparison: Belzutifan vs Everolimus; Test type: Superiority; p = 0.00031, Log Rank; One-sided p-value based on log-rank test stratified by IMDC Risk Category and Number of prior VEGF/VEGF-Receptor Targeted Therapies for RCC; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.63 to 0.88] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by IMDC Risk Category and Number of prior VEGF/VEGF-Receptor Targeted Therapies for RCC

2. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up.
Time Frame: Up to approximately 49 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belzutifan | Everolimus
Number analyzed (Participants) | 374 | 372
Months | 21.4 [18.2 to 24.3] | 18.2 [15.8 to 21.8]
Statistical Analysis 1: Comparison: Belzutifan vs Everolimus; Test type: Superiority; p = 0.17644, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.77 to 1.10] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by BICR
Description: ORR is defined as the percentage of participants who have a complete response (CR: Disappearance of all target lesions) or a partial response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience a CR or PR as assessed by blinded independent central review based on RECIST 1.1 is presented here.
Time Frame: Up to approximately 31 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Belzutifan | Everolimus
Number analyzed (Participants) | 374 | 372
Percentage of Participants | 21.9 [17.8 to 26.5] | 3.5 [1.9 to 5.9]
Statistical Analysis 1: Comparison: Belzutifan vs Everolimus; Test type: Superiority — P-value, difference in percentage and associated 95% CI were calculated using Miettinen & Nurminen method stratified by IMDC Risk Category and Number of prior VEGF/VEGF-Receptor Targeted Therapies for RCC; p < 0.00001, Miettinen & Nurminen — One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = 18.4, 95% CI 2-sided [14.0 to 23.2] — Belzutifan minus Everolimus

4. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR
Description: For participants who demonstrate a confirmed complete response (CR: Disappearance of all target lesions) or confirmed partial response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death. The DOR as assessed by blinded independent central review is presented here. The Median DOR was analyzed by the Kaplan-Meier method for censored data.
Time Frame: Up to approximately 49 months
Population: Per protocol, the analysis population consisted of all randomized participants based on the treatment group to which they were randomized, and who experienced a confirmed complete response (CR) or partial response (PR). Per protocol, participants enrolled in the Safety Run-In were not randomized and not included in the protocol-specified analyses for any of the outcome measures.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belzutifan | Everolimus
Number analyzed (Participants) | 85 | 13
Months | 19.3 [14.0 to 28.6] | 13.7 [5.6 to 20.5]

5. Secondary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs)
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to approximately 78 months
Reporting Status: Not Posted

6. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of participants who discontinue study treatment due to an AE will be presented.
Time Frame: Up to approximately 78 months
Reporting Status: Not Posted

7. Secondary Outcome: Time to True Deterioration (TTD) in Health-Related Quality-of-Life (HRQoL) Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Items 29 and 30 Combined Score
Description: The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to the questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and Quality of Life (QoL; "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent), then summed. Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. TTD was defined as the time from baseline to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in Items 29 and 30 scale scores. If the first deterioration is at the last PRO assessment timepoint at the time of analysis, then no confirmation is required. A longer TTD indicates a better outcome. TTD is reported based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 39 months
Population: Per protocol, the analysis population consisted of all randomized participants who have at least one assessment available for EORTC QLQ-C30 and have received at least one dose of the study intervention; and had data available for this TTD in HRQoL outcome using EORTC QLQ-C30. Per protocol, participants enrolled in the Safety Run-In were not randomized and not included in the protocol-specified analyses for any of the outcome measures.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belzutifan | Everolimus
Number analyzed (Participants) | 351 | 333
Months | 19.35 [11.89 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 10.19 [6.47 to 12.98]
Statistical Analysis 1: Comparison: Belzutifan vs Everolimus; Test type: Other; p = 0.0185, Log Rank; Two-sided p-value based on log-rank test stratified by IMDC Risk Category and Number of prior VEGF/VEGF-Receptor Targeted Therapies for RCC; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.58 to 0.96] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: TTD in Physical Functioning Using the EORTC QLQ-C30 Items 1- 5 Score
Description: The EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much), then summed. Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. TTD was defined as the time from baseline to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in physical functioning Items 1 to 5 scale scores. If the first deterioration is at the last PRO assessment timepoint at the time of analysis, then no confirmation is required. A longer TTD indicates a better outcome. TTD is reported based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 39 months
Population: Per protocol, the analysis population consisted of all randomized participants who have at least one assessment available for EORTC QLQ-C30 and have received at least one dose of the study intervention; and had data available for this TTD in physical functioning outcome using EORTC QLQ-C30. Per protocol, participants enrolled in the Safety Run-In were not randomized and not included in the protocol-specified analyses for any of the outcome measures.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belzutifan | Everolimus
Number analyzed (Participants) | 351 | 333
Months | 19.32 [11.11 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 13.83 [10.61 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Belzutifan vs Everolimus; Test type: Other; p = 0.5533, Log Rank; [statistical method as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.72 to 1.20] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: TTD in Disease Symptoms Using the Functional Assessment of Cancer Therapy-Kidney Symptom Index-Disease-related Symptoms (FKSI-DRS) Items 1-9 Score
Description: The FKSI-DRS was a questionnaire that asked the participant to rate 9 kidney cancer-related symptoms: lack of energy, fatigue, weight loss, pain, bone pain, shortness of breath, cough, fever, or blood in the urine. Each item was scored on a 5-point scale (0=not at all to 4=very much). FKSI-DRS total score ranged from 0 (most severe symptoms) to 36 (no symptoms) with a higher score indicating a better outcome. TTD was defined as the time to first onset of a ≥3-point decrease in symptom score from baseline with confirmation by the subsequent visit of a ≥3-point deterioration from baseline under right-censoring rule. If the first deterioration is at the last PRO assessment timepoint at the time of analysis, then no confirmation is required. A longer TTD indicates a better outcome. TTD is reported based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 39 months
Population: Per protocol, the analysis population consisted of all randomized participants who have at least one assessment available for FKSI-DRS and have received at least one dose of the study intervention; and had data available for this TTD in disease symptoms outcome using FKSI-DRS. Per protocol, participants enrolled in the Safety Run-In were not randomized and not included in the protocol-specified analyses for any of the outcome measures.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belzutifan | Everolimus
Number analyzed (Participants) | 352 | 334
Months | NA [21.26 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 11.99 [5.55 to 15.38]
Statistical Analysis 1: Comparison: Belzutifan vs Everolimus; Test type: Other; p < 0.0001, Log Rank; [statistical method as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.41 to 0.69] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change From Baseline to Week 17 in the HRQoL Using the EORTC QLQ-C30 Items 29 and 30 Combined Score
Description: The EORTC-QLQ-C30 is a 30-item questionnaire to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the Quality of Life (QoL) question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100; a higher score indicating a better overall outcome. Change from baseline to Week 17 in EORTC QLQ-C30 Items 29 and 30 combined scores was calculated based on a constrained longitudinal data analysis (cLDA) model with scores as response variable with covariates for treatment by time interaction, stratification factors (IMDC Risk Category, and Number of Prior VEGF/VEGF-Receptor Targeted Therapies for RCC) as covariates.
Time Frame: Baseline (Day 1) and week 17
Population: Per protocol, the analysis population consisted of all randomized participants who have received at least one dose of the study intervention and had assessments available for EORTC QLQ-C30 at baseline or post-baseline up to Week 17; and had data available for this change from baseline in HRQoL outcome using EORTC QLQ-C30. Per protocol, participants enrolled in the Safety Run-In were not randomized and not included in the protocol-specified analyses for any of the outcome measures.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Belzutifan | Everolimus
Number analyzed (Participants) | 363 | 353
Score on a Scale | 0.28 [-1.98 to 2.53] | -6.11 [-8.51 to -3.70]
Statistical Analysis 1: Comparison: Belzutifan vs Everolimus; Test type: Other; p < 0.0001, t-test, 2 sided; Difference in Least Squares (LS) Means = 6.38, 95% CI 2-sided [3.21 to 9.55] — Based on a cLDA model with scores as the response variable with covariates for treatment by time interaction, stratification factors (IMDC Risk Category, and Number of Prior VEGF/VEGF-Receptor Targeted Therapies for RCC) as covariates

11. Secondary Outcome: Change From Baseline to Week 17 in Physical Functioning Using the EORTC QLQ-C30 Items 1- 5 Score
Description: The EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much), then summed. Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. The change from baseline to Week 17 in physical functioning (EORTC QLQ-C30 Items 1-5) score was calculated based on a constrained longitudinal data analysis (cLDA) model with scores as response variable with covariates for treatment by time interaction, stratification factors (IMDC Risk Category, and Number of Prior VEGF/VEGF-Receptor Targeted Therapies for RCC) as covariates.
Time Frame: Baseline (Day 1) and week 17
Population: Per protocol, the analysis population consisted of all randomized participants who have received at least one dose of the study intervention and had assessments available for EORTC QLQ-C30 at baseline or post-baseline up to Week 17; and had data available for this change from baseline in physical functioning outcome using EORTC QLQ-C30. Per protocol, participants enrolled in the Safety Run-In were not randomized and not included in the protocol-specified analyses for any of the outcome measures.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Belzutifan | Everolimus
Number analyzed (Participants) | 363 | 353
Score on a Scale | -4.75 [-6.87 to -2.63] | -7.22 [-9.47 to -4.98]
Statistical Analysis 1: Comparison: Belzutifan vs Everolimus; Test type: Other; p = 0.1134, t-test, 2 sided; Difference in LS Means = 2.47, 95% CI 2-sided [-0.59 to 5.54] — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Change From Baseline to Week 17 in Disease Symptoms Using the FKSI-DRS Items 1-9 Score
Description: The FKSI-DRS was a questionnaire that asked the participant to rate 9 kidney cancer-related symptoms: lack of energy, fatigue, weight loss, pain, bone pain, shortness of breath, cough, fever, or blood in the urine. Each item was scored on a 5-point scale (0=not at all to 4=very much). FKSI-DRS total score ranged from 0 (most severe symptoms) to 36 (no symptoms) with a higher score indicating a better outcome. The change from baseline to Week 17 in Disease Symptoms using the FKSI-DRS Items 1-9 score was calculated based on a constrained longitudinal data analysis (cLDA) model with the PRO scores as response variable with covariates for treatment by time interaction, stratification factors (IMDC Risk Category, and Number of Prior VEGF/VEGF-Receptor Targeted Therapies for RCC) as covariates.
Time Frame: Baseline (Day 1) and week 17
Population: Per protocol, the analysis population consisted of all randomized participants who have received at least one dose of the study intervention and had assessments available for FKSI-DRS at baseline or post-baseline up to Week 17; and had data available for this change from baseline in disease symptoms outcome using FKSI-DRS. Per protocol, participants enrolled in the Safety Run-In were not randomized and not included in the protocol-specified analyses for any of the outcome measures.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Belzutifan | Everolimus
Number analyzed (Participants) | 363 | 353
Score on a Scale | -0.17 [-0.70 to 0.36] | -1.62 [-2.17 to -1.06]
Statistical Analysis 1: Comparison: Belzutifan vs Everolimus; Test type: Other; p = 0.0002, t-test, 2 sided; Difference in LS Means = 1.45, 95% CI 2-sided [0.70 to 2.19] — Based on a cLDA model with the PRO scores as the response variable with covariates for treatment by time interaction, stratification factors (IMDC Risk Category, and Number of Prior VEGF/VEGF-Receptor Targeted Therapies for RCC) as covariates

13. Secondary Outcome: Change From Baseline to Week 17 in Visual Analogue Scale (VAS) Score on the European Quality of Life 5 Dimension, 5-level Questionnaire (EQ-5D-5L) Health Utility Score
Description: The EQ-5D-5L questionnaire assesses 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/ depression. Each dimension has 5 response options that reflect increasing levels of difficulty, which are coded on a scale from 1 (no problems) to 5 (extreme problems). The VAS is a component of EQ-5D-5L that asks participants to rate their overall health on a vertical visual analogue scale, with the scale's ends labelled 'The best health you can imagine' (equivalent to a score of 0) and 'The worst health you can imagine' (equivalent to a score of 100). The change from baseline to Week 17 in Health Utility using the EQ-5D-5L VAS score was calculated based on a constrained longitudinal data analysis (cLDA) model with the PRO scores as response variable with covariates for treatment by time interaction, stratification factors (IMDC Risk Category, and Number of Prior VEGF/VEGF-Receptor Targeted Therapies for RCC) as covariates.
Time Frame: Baseline (Day 1) and week 17
Population: Per protocol, the analysis population consisted of all randomized participants who have received at least one dose of the study intervention with assessments available for EQ-5D-5L at baseline or post-baseline up to Week 17; and had data available in this change from baseline in VAS Score using EQ-5D-5L. Per protocol, participants enrolled in the Safety Run-In were not randomized and not included in the protocol-specified analyses for any of the outcome measures.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Belzutifan | Everolimus
Number analyzed (Participants) | 363 | 353
Score on a Scale | -0.19 [-2.03 to 1.65] | -3.91 [-5.86 to -1.96]
Statistical Analysis 1: Comparison: Belzutifan vs Everolimus; Test type: Other; p = 0.0051, t-test, 2 sided; Difference in LS Means = 3.72, 95% CI 2-sided [1.12 to 6.31] — [estimate comment as in outcome 12, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to approximately 49 months
Description: Serious and Other adverse events (AEs) include all participants who received ≥1 dose of study drug. All-Cause Mortality includes all enrolled participants. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Groups:
- Belzutifan: Randomized participants receive 120 mg of belzutifan orally once daily (QD), until disease progression or discontinuation.
- Everolimus: Randomized participants receive 10 mg of Everolimus orally QD, until disease progression or discontinuation.
Arm/Group | Belzutifan | Everolimus | Safety Run-In
All-Cause Mortality (participants affected / at risk) | 254/374 | 259/372 | 5/9
Serious Adverse Events (participants affected / at risk) | 160/372 | 139/360 | 4/9
Other Adverse Events (participants affected / at risk) | 356/372 | 348/360 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belzutifan (N=372) | Everolimus (N=360) | Safety Run-In (N=9)
Anaemia (Blood and lymphatic system disorders) | 20 (21) | 8 (8) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 4 (5) | 5 (5) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 3 (4) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Cystoid macular oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fistula of small intestine (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 3 (3) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hernia pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 4 (4) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 9 (9) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 5 (5) | 11 (11) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 18 (21) | 17 (17) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Prostatitis Escherichia coli (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (2) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral pericarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Shoulder fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Resorption bone increased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 6 (6) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (4) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 27 (29) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 10 (13) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 16 (16) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Assisted suicide (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Belzutifan (N=372) | Everolimus (N=360) | Safety Run-In (N=9)
Anaemia (Blood and lymphatic system disorders) | 294 (503) | 200 (272) | 8 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (23) | 25 (34) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 29 (38) | 21 (23) | 0 (0)
Constipation (Gastrointestinal disorders) | 63 (78) | 30 (30) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 47 (63) | 71 (87) | 0 (0)
Nausea (Gastrointestinal disorders) | 68 (96) | 44 (46) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 13 (15) | 137 (173) | 0 (0)
Vomiting (Gastrointestinal disorders) | 47 (62) | 31 (32) | 2 (2)
Asthenia (General disorders) | 55 (67) | 60 (63) | 0 (0)
Chest pain (General disorders) | 20 (21) | 10 (10) | 0 (0)
Fatigue (General disorders) | 120 (138) | 91 (100) | 2 (2)
Oedema peripheral (General disorders) | 64 (74) | 65 (71) | 1 (1)
Pyrexia (General disorders) | 20 (23) | 43 (64) | 2 (2)
COVID-19 (Infections and infestations) | 37 (39) | 25 (32) | 0 (0)
Pneumonia (Infections and infestations) | 7 (8) | 19 (20) | 0 (0)
Urinary tract infection (Infections and infestations) | 20 (29) | 20 (27) | 0 (0)
Alanine aminotransferase increased (Investigations) | 47 (64) | 33 (38) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 42 (61) | 33 (43) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 19 (22) | 21 (24) | 0 (0)
Blood creatinine increased (Investigations) | 32 (47) | 43 (52) | 2 (2)
Blood triglycerides increased (Investigations) | 17 (24) | 22 (27) | 0 (0)
Platelet count decreased (Investigations) | 13 (16) | 19 (30) | 2 (2)
Weight decreased (Investigations) | 15 (15) | 33 (34) | 0 (0)
Weight increased (Investigations) | 22 (29) | 2 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 54 (59) | 57 (61) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (14) | 54 (69) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 15 (26) | 53 (65) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (6) | 19 (32) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 19 (30) | 12 (15) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 60 (72) | 29 (33) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 61 (74) | 31 (33) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 21 (25) | 13 (17) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 (35) | 25 (26) | 0 (0)
Dizziness (Nervous system disorders) | 50 (73) | 6 (9) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3) | 23 (23) | 0 (0)
Headache (Nervous system disorders) | 48 (58) | 28 (30) | 0 (0)
Insomnia (Psychiatric disorders) | 22 (24) | 19 (22) | 1 (1)
Proteinuria (Renal and urinary disorders) | 10 (15) | 21 (22) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (37) | 76 (82) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 55 (69) | 46 (49) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 29 (34) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 29 (41) | 4 (4) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 39 (42) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 31 (34) | 59 (62) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 17 (17) | 69 (78) | 0 (0)
Hypertension (Vascular disorders) | 26 (28) | 25 (30) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1) | 4 (4) | 2 (2)
Macular oedema (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 9 (11) | 7 (8) | 1 (1)
Malaise (General disorders) | 8 (9) | 2 (2) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 3 (3) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 3 (3) | 3 (3) | 1 (1)
Herpes zoster (Infections and infestations) | 13 (14) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 8 (10) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 4 (5) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (5) | 6 (8) | 1 (1)
White blood cell count decreased (Investigations) | 2 (2) | 11 (17) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0/9 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (6) | 16 (18) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT04195750/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT04195750/SAP_001.pdf